CLINICAL TRIAL: NCT07362940
Title: A Phase Ⅰ/Ⅱa Clinical Study Evaluating the Efficacy and Safety of GEN-725 in Combination With Dositinib in Patients With Locally Advanced or Metastatic EGFR-Mutant Non-small Cell Lung Cancer
Brief Title: A Phase Ⅰ/Ⅱa Clinical Study of GEN-725 in Combination With Dositinib
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Dox-RC001
Record Dates: First submitted 2025-12-24; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; EGFR mutation; GEN -725; Dositinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Dose-escalation part and dose-expansion part
  Interventions: Drug: GEN-725 tablets + Dositinib mesylate tablets

INTERVENTIONS:
Drug: GEN-725 tablets + Dositinib mesylate tablets — Dose-escalation part (Phase Ⅰ): Subjects will receive once-daily oral administration of GEN-725 tablets in combination with Dositinib mesylate tablets on an empty stomach. GEN-725 will be administered at a dose of 6 mg or 9 mg, and Dositinib will be administered at a dose of 80 mg or 160 mg. Both drugs should be taken concurrently. The treatment will continue until the first occurrence of any of the following: disease progression, unacceptable toxicity, withdrawal of consent, or investigator's determination of no further clinical benefit.
  Dose-expansion part (Phase Ⅱa): Subjects will receive once-daily oral administration of GEN-725 tablets in combination with Dositinib mesylate tablets or Dositinib mesylate tablets alone on an empty stomach. The dose will be selected based on the outcome of dose-escalation phase. The treatment will continue until the first occurrence of any criterion that was specified in the dose-escalation part.

SUMMARY:
This is an open-label phase I/phase II clinical study designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of GEN-725 in combination with Dositinib in participants with locally advanced or metastatic EGFR-mutant non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old (including 18 and 75 years old), male or female.
2. Patients with histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) who are not amenable to curative surgery or radiotherapy. (For subjects naive to EGFR-TKI therapy, paraffin-embedded tissue blocks, unstained slides, or fresh tumor tissue samples must be available for EGFR testing.)
3. Patients with a positive EGFR mutation. (For patients with prior third-generation EGFR-TKI therapy, post-progression EGFR mutation test results are recommended.)
4. a) Phase Ⅰ Dose Escalation Stage: EGFR-mutant NSCLC patients who have received at least one prior line of therapy (chemotherapy or targeted therapy are allowed). Patients who have received prior neoadjuvant, adjuvant, and/or radical concurrent/sequential chemoradiotherapy (including chemotherapy, immunotherapy, targeted therapy, etc.) must have documented disease recurrence or progression within <6 months of completing the last regimen. b) Phase Ⅱa Dose Expansion Stage: Cohort 1: NSCLC patients with disease progression on a prior third-generation EGFR-TKI. Cohort 2: EGFR mutant NSCLC patients who are EGFR-TKI-naive.
5. Patients with at least one measurable or evaluable lesion per RECIST 1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and a life expectancy of at least 12 weeks.
7. Adequate organ function must meet the following criteria (with no transfusion of blood, blood products, no administration of hematopoietic growth factors, or no infusion of albumin/blood products within 14 days before laboratory testing):

   1. Absolute neutrophil (NE) count ≥ 1.5 × 10^9/L.
   2. Platelet (PLT) count ≥ 100 × 10^9/L.
   3. Hemoglobin (HGB) ≥ 100 g/L.
   4. Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 × ULN (for patients with liver metastases, TBIL ≤ 3 × ULN and AST/ALT ≤ 5 × ULN are acceptable).
   5. Serum creatinine (SCr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min. Note: If the investigator deems retesting necessary (with the reason documented), the above laboratory tests may be repeated only once. If the retesting results meet the criteria, they will be considered eligible.
8. Patients with stable intracranial metastatic lesions are eligible. Stable intracranial metastasis is defined as: stable signs and symptoms for at least 2 weeks before enrollment, and discontinuation of corticosteroid treatment for intracranial metastasis for at least 14 days before enrollment. Patients with stable intracranial metastases (including newly identified intracranial metastasis that are treatment-naive) who do not require treatment are eligible. Patients with stable meningeal metastasis are eligible following confirmation by the investigator (Applicable only to dose expansion stage).
9. Women of childbearing potential must have a negative blood pregnancy test and agree to use effective contraception during the study treatment and for 180 days after the last administration. According to the judgment of the investigator, women of childbearing potential in this study are defined as sexually mature women: 1) have not undergone a hysterectomy or bilateral oophorectomy; 2) have not experienced natural menopause last for 12 consecutive months (amenorrhea following cancer treatment does not preclude the possibility of fertility) (i.e., have experienced menstruation with the last 12 consecutive months). Male patients with female partners of childbearing potential must agree to use effective contraception during the study treatment and for 180 days after the last administration.
10. Subjects have been fully informed, have voluntarily sign the informed consent form, and are willing to comply with the study procedures and visit schedule.

Exclusion Criteria:

1. Patients have previously received any of the following treatments:

   1. Undergone major surgery within 4 weeks prior to the first administration;
   2. Antitumor therapy including chemotherapy, immunotherapy, targeted therapy, etc., within 4 weeks prior to the first administration; for oral small-molecule targeted drugs, within 2 weeks or within 5 half-lives prior to the first administration (whichever is shorter);
   3. Radiation therapy involving >30% of the bone marrow or large-field radiation therapy within 4 weeks prior to the first administration;
   4. Strong inhibitors or inducers of CYP3A4 within 7 days prior to the first administration;
   5. Traditional Chinese medicine (TCM) or TCM preparations that have antitumor indications, or that are intended for tumor adjuvant therapy within 14 days prior to the first administration;
2. Presence of unresolved toxicities from previous anticancer therapy, with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade >1 (except alopecia) at the start of study treatment. The pre-existing neuropathy from previous platinum-therapy is allowed up to grade 2;
3. Patients with meaningful bypass mutations of corresponding marketed drugs, including but not limited to: MET exon 14 skipping mutation, MET amplification, ALK fusion, HER-2 mutation, ROS-1 fusion, RET fusion, BRAF V600E mutation, KRAS G12C, NTRK fusion, etc. (Applicable only to the dose expansion period, and will be adjusted according to the gene detection results from the dose escalation period);
4. Patients with disease progression (PD) or stable disease (SD) with a duration of ≤3 months following treatment with a third-generation EGFR-TKI;
5. Patients with any uncontrolled systemic disease, as determined by the investigator, such as uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg after optimal medical therapy), uncontrolled diabetes, coronary artery stenosis, aortic dissection, aortic aneurysm, active bleeding diathesis, etc.;
6. Patients with any clinically significant gastrointestinal condition that could impair the intake, transport, or absorption of the study drug, such as inability to take oral medication, uncontrollable nausea and vomiting, history of major gastrointestinal resection, uncured chronic diarrhea, atrophic gastritis (age of onset <60 years), uncured gastric diseases requiring long-term use of proton pump inhibitors (e.g., omeprazole, lansoprazole, pantoprazole, rabeprazole), Crohn's disease, ulcerative colitis, etc.;
7. Patients meeting any of the following cardiac criteria:

   1. Mean corrected QT interval (QTc) >470 msec based on resting electrocardiogram (ECG);
   2. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG, such as complete left bundle branch block, Ⅲ degree atrioventricular block, Ⅱ degree atrioventricular block, or PR interval >250 msec, etc.;
   3. Congestive heart failure classified as New York Heart Association (NYHA) Class III-IV, or poorly controlled and clinically significant arrhythmias;
   4. Any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome in first-degree relatives or unexplained sudden death under 40 years of age, or current use of any medication known to prolong the QT interval;
8. Left ventricular ejection fraction (LVEF) <50% as measured by echocardiography;
9. Patients with interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid treatment; or those with suspected ILD/non-infectious pneumonitis that cannot be ruled out by imaging during screening;
10. Patients with concurrent pulmonary disease resulting in clinically severe respiratory impairment, including but not limited to: severe pulmonary embolism within 3 months prior to the first dose, severe asthma, or severe chronic obstructive pulmonary disease, etc.;
11. Patients with a history of significant arterial/venous thrombotic events or cerebrovascular accidents within 6 months prior to the first administration, such as pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc.; with the exception of asymptomatic lacunar infarction or intramuscular venous thrombosis not requiring clinical intervention;
12. Patients with concurrent use of therapeutic doses of anticoagulants such as vitamin K antagonists or heparin (patients using prophylactic doses are eligible);
13. Patients with an active systemic infection: Tuberculosis (clinical diagnosis including history, physical examination, radiographic findings, and TB testing per local practice), Hepatitis B (HBsAg positive and HBV DNA ≥500 copies/ml or above the upper limit of the normal reference range), Hepatitis C (HCV RNA above the upper limit of normal), or Human Immunodeficiency Virus (HIV antibody positive);
14. Patients with clinically uncontrolled pleural effusion/ascites/pericardial effusion within 2 weeks prior to the first administration. (Patients are eligible if the effusion does not require drainage or has shown no significant increase for 3 days after drainage cessation);
15. Patients with a history of other malignancies within 5 years prior to the first administration, except for: adequately treated papillary thyroid carcinoma, basal cell or squamous cell skin cancer, or other in situ carcinomas that have been adequately treated with no evidence of recurrence (including but not limited to cervical carcinoma in situ, ductal carcinoma in situ of the breast, etc.);
16. Patients who have received systemic corticosteroids (>10 mg/day prednisone equivalent) or other systemic immunosuppressants (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents) within 2 weeks prior to the first administration. The use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroids is permitted;
17. Patients with a history of psychiatric disorders or substance abuse that may impair compliance with trial requirements;
18. Patients with a history of other acquired or congenital immunodeficiency diseases, or those who have undergone or are scheduled for organ transplantation or bone marrow transplantation;
19. Patients with a history of hypersensitivity to the active ingredient or any excipients of the study drug, or to any drug of a similar chemical structures or pharmacological class;
20. Patients with any other acute or chronic medical conditions, psychiatric conditions, or abnormal laboratory findings that may increase the risk associated with study participation or study drug administration, or interfere with result interpretation, and, in the investigator's judgment, make the patients unsuitable for participation in this study;
21. Patients who are unlikely to comply with the study protocol, or in the investigator's opinion, the patient is unsuitable for participation in this clinical study due to other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Dose Limiting Toxicity (DLT) in Phase Ⅰ | From Day 1 to Day 21 of Cycle1 (each cycle is 21 days).
Incidence and severity of adverse events (AEs) in Phase Ⅰ and Phase Ⅱa | From the time of informed consent until 28 days after the last administration of the study drugs.
  AEs are assessed based on NCI CTCAE v5.0.
Objective Response Rate (ORR) in Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Intracranial Objective Response Rate (iORR) in Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in Phase Ⅰ | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Disease Control Rate (DCR) in Phase Ⅰ and Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Progression-Free Survival (PFS) in Phase Ⅰ and Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Duration of Response (DOR) in Phase Ⅰ and Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Overall Survival (OS) in Phase Ⅰ and Phase Ⅱa | Every 12 weeks after the last dose, up to 5 years, up to 5 years.
Intracranial Progression-Free Survival (iPFS) in Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Intracranial Disease Control Rate (iDCR) in Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Intracranial Duration of Response (iDOR) in Phase Ⅱa | Every 6 weeks during the first year and every 12 weeks thereafter, up to 5 years.
Maximum Plasma Concentration (Cmax) of GEN-725 and Dositinib | Up to 24 hours post-dose.
Elimination Half-Life (t1/2) of GEN-725 and Dositinib | Up to 24 hours post-dose.
Area Under the Plasma Concentration Curve (AUC) of GEN-725 and Dositinib | Up to 24 hours post-dose.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Cancer Hospital Affiliated to Shandong First Medical University (Shandong Cancer Hospital, Shandong cancer prevention and treatment institute), Jinan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou